CLINICAL TRIAL: NCT07149051
Title: Design and Implementation of a Gamified Sensory Integration Exercise Intervention
Brief Title: Design of a Sensory Integration Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof., Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEE2055
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Sensory Integration Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention program consists of gamified physical activities, incorporating game elements such as game scenarios, mechanisms, and components into the teaching content.
  Interventions: Behavioral: Gamified Sensory Integration Exercise Program
- Control Group (No Intervention): Participants in the control group received the regular physical education curriculum.

INTERVENTIONS:
Behavioral: Gamified Sensory Integration Exercise Program — This study implemented a gamified physical activity intervention aimed at improving sensory integration abilities among first-grade students with sensory processing difficulties. The intervention program incorporated game narratives, mechanisms, and components into physical education activities, guided by the Octalysis Framework to strategically engage both extrinsic (e.g., rewards, rankings) and intrinsic (e.g., creativity, social interaction, meaning) motivational drives.
  Arms: Intervention Group

SUMMARY:
This study aims to explore the mechanisms of motor skill promotion and sensory integration intervention for first-grade primary school students with sensory integration dysfunction. By designing a gamified exercise intervention program tailored to lower-grade students, and combining it with the assessment and analysis of sensory integration functions, the study seeks to systematically improve their sensory integration ability and physical fitness, thereby supporting healthy growth and enhanced adaptability during this critical stage of physical and psychological development.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 7 years;
* Diagnosis of sensory integration dysfunction in at least one subscale of the assessment tool;
* Informed consent was obtained from both legal guardians and teachers.

Exclusion Criteria:

* Physical deformities or other conditions limiting participation in physical activities;
* Serious medical conditions;
* Severe cognitive impairments that could interfere with comprehension or participation in the intervention.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Sensory Integration Ability | Month 3
  Sensory integration ability was measured using the Participants' Sensory Integration Development Evaluation Scale. The scale consists of 58 items rated on a five-point Likert scale and covers vestibular function, tactile defensiveness, proprioception, learning ability, and special problems; the last dimension was excluded due to the participants' age. Assessments were conducted at baseline and at three months.
Speed Test | Month 3
  was measured using the 50 m sprint. Assessments were conducted at baseline and at three months.
Flexibility Test | Month 3
  Flexibility was measured using the sit-and-reach test. Assessments were conducted at baseline and at three months.
Coordination Test | Month 3
  Coordination was measured using the one-minute rope skipping test. Assessments were conducted at baseline and at three months.
Balance Test | Month 3
  Balance was measured using the single-leg stance with eyes closed. Assessments were conducted at baseline and at three months.
Lower-limb strength Test | Month 3
  Lower-limb strength was measured using the standing long jump. Assessments were conducted at baseline and at three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No